CLINICAL TRIAL: NCT00042848
Title: Phase III Randomized, Placebo-Controlled, Double-Blind Trial Of The Effect Of Modafinil On Fatigue In Cancer Patients Receiving Chemotherapy
Brief Title: Modafinil in Treating Fatigue in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000069477; U10CA037420 (NIH); URCC-U2901 (Other: University of Rochester)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Fatigue | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: modafinil

SUMMARY:
RATIONALE: Modafinil may be effective in relieving fatigue in patients with cancer who are undergoing chemotherapy. The effectiveness of modafinil in relieving chemotherapy-related fatigue is not yet known.

PURPOSE: This randomized phase III trial is studying the effectiveness of modafinil in treating fatigue in patients who are receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the degree to which modafinil can reduce fatigue in cancer patients receiving chemotherapy.
* Assess the relationship between depression and fatigue in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on day 5 of the second course of chemotherapy, patients receive oral modafinil once daily.
* Arm II: Beginning on day 5 of the second course of chemotherapy, patients receive oral placebo once daily.

Treatment in both arms continues until day 7 of course 4 of chemotherapy in the absence of disease progression or unacceptable toxicity.

Fatigue and quality of life are assessed on day 7 of courses 2-4 of chemotherapy.

PROJECTED ACCRUAL: A total of 837 patients will be accrued for this study within approximately 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Concurrently receiving or has previously received chemotherapy and is scheduled for at least 3 additional courses of chemotherapy

  * Each course of chemotherapy must be at least 2 weeks in duration
  * No concurrent radiotherapy or interferon therapy
* Brief Fatigue Inventory question #3 "fatigue worst" score of 2 or greater 1 week after first chemotherapy course

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* No uncontrolled anemia

Renal

* Not specified

Cardiovascular

* No history of clinically significant cardiac disease, including any of the following:

  * Unstable angina
  * Left ventricular hypertrophy
  * Ischemic echocardiogram changes
  * Chest pain
  * Arrhythmia
  * Other clinically significant manifestations of mitral valve prolapse in association with use of central nervous system stimulants (e.g., caffeine, amphetamines, or methylphenidate)
* No uncontrolled hypertension

Gastrointestinal

* Able to swallow medication
* No narrowing (pathological or iatrogenic) or obstruction of the gastrointestinal tract

Other

* No severe headaches
* No glaucoma
* No seizure disorder
* No narcolepsy
* No psychotic disorder
* No Tourette's syndrome
* No alcohol or drug abuse
* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for at least 1 full menstrual cycle after study completion

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* No concurrent chronic corticosteroids

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Other

* No prior modafinil
* At least 30 days since prior regular use of psychostimulants (e.g., amphetamines, methylphenidate, or pemoline) or monoamine oxidase inhibitors (MAOIs)
* No concurrent alcohol
* Concurrent acetaminophen with codeine or hydrocodone bitartrate allowed
* Concurrent phenytoin allowed
* Concurrent warfarin for anticoagulation and low-dose warfarin (1 mg by mouth daily) for maintenance of venous access devices allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Efficacy to reduce fatigue during chemotherapy as assessed by the Brief Fatigue Inventory at course 4

SECONDARY OUTCOMES:
Relationship between depression and fatigue during chemotherapy as assessed by Fatigue Symptom Checklist, Profile of Mood States, Fatigue Severity Scale, Epworth Sleepiness Scale, Center for Epidemiologic Studies-Depression, and Mini-Mac at course 4

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — James P. Wilmot Cancer Center
Locations (35):
- United States (35):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Denver Rose, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers - Longmont, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Jean-Pierre P, Morrow GR, Roscoe JA, Heckler C, Mohile S, Janelsins M, Peppone L, Hemstad A, Esparaz BT, Hopkins JO. A phase 3 randomized, placebo-controlled, double-blind, clinical trial of the effect of modafinil on cancer-related fatigue among 631 patients receiving chemotherapy: a University of Rochester Cancer Center Community Clinical Oncology Program Research base study. Cancer. 2010 Jul 15;116(14):3513-20. doi: 10.1002/cncr.25083. PMID 20564068